CLINICAL TRIAL: NCT04759339
Title: An Open Label, Non-Comparative Study of the Systemic Exposure to Articaine After Topical Ocular Dosing of Articaine Sterile Topical Ophthalmic Solution (AG-920)
Brief Title: An Open Label, Study of the Systemic Exposure to Articaine After Topical Ocular Dosing of AG-920
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Genomics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AG-920-CS101
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: articaine; AG-920

STUDY DESIGN:
Intervention Model Description: An open label, non-comparative study of the systemic exposure to articaine after topical ocular dosing of articaine sterile topical ophthalmic solution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG-920 (Experimental): Subjects will receive a single dose of articaine sterile topical ophthalmic solution in one eye only. The study eye will be randomized. The single dose will be administered by the clinic staff as two drops in study eye 30 seconds apart.
  Interventions: Drug: AG-920

INTERVENTIONS:
Drug: AG-920 — AG-920 is a sterile, isotonic, non-preserved aqueous solution containing the active ingredient Articaine HCl 8%
  Other Names: Articaine Sterile Topical Ophthalmic Solution

SUMMARY:
This is a Phase 1, open-label, non-comparative study in healthy subjects performed in the US. It is designed to assess systemic exposure to articaine and its metabolite articainic acid after dosing a single topical ocular administration of AG-920 in the randomized study eye.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-comparative study in healthy subjects designed to assess systemic exposure to articaine and its metabolite articainic acid after dosing a single topical ocular administration of AG-920 in the randomized study eye.

In this study, subjects who provide informed consent and fulfill all the inclusion criteria and none of the exclusion criteria will receive a single dose of study drug in one eye. The study eye will be randomized. The single dose will be administered by the clinic staff as two drops 30 seconds apart in study eye. Subjects will have pharmacokinetic (PK) blood samples taken at multiple periods over 24 hours following dosing. Safety will be assessed by monitoring any changes in heart rate, blood pressure, intraocular pressure, visual acuity, biomicroscopy, and AEs.

The study will consist of 3 clinical visits: Screening Visit, Dosing and PK Blood Level Sampling (0-8 hours) Visit and a Follow Up Visit (with PK blood level sampling 24 hours after study drug treatment).

ELIGIBILITY:
Key Inclusion Criteria:

1. Voluntarily provide written informed consent prior to any study-related procedures being performed.
2. Female subjects of childbearing potential must have negative pregnancy test.
3. Certified as healthy by clinical assessment.
4. Have an Early Treatment of Diabetic Retinopathy Study best corrected visual acuity of 20/200 or better in each eye.
5. Have an Intraocular Pressure between 7 and 30 mmHg inclusive.
6. Are able to tolerate instillation of Over-The-Counter artificial tear product .
7. Blood pressure < 140/90 mmHg and heart rate < 100 bpm at screening.

Key Exclusion Criteria:

1. Have previously received AG-920.
2. Have a contraindication to local anesthetics.
3. Have had ocular surgery or general surgery within the past 90 days.
4. Have had an intravitreal injection in either eye within 14 days of treatment.
5. Have a history within the last year of or current ocular surface disease or nasolacrimal duct abnormalities including obstructions or requiring punctal plugs.
6. Have evidence of any current ocular inflammation.
7. Have a known current condition which could cause vision problems.
8. Current ocular allergy symptoms.
9. Have donated or lost more than 400 mL of blood within 12 weeks.
10. Plasma donation within 7 days prior to the first dosing.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Systemic exposure to articaine and its metabolite after dosing a single topical ocular administration of AG-920 | 8 hours
  Plasma levels of articaine and its primary metabolite (articainic acid)

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAE) | randomization through follow up (2 days)
  TEAEs will be summarized by system organ class (SOC) and preferred term.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Uram, MD, Study Director — American Genomics, LLC
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verhoeven R, Uram M, Schupp A, Rasmussen S, Widmann M, Novack GD. Early Nonclinical and Clinical Development of AG-920, a Repurposed Topical Ocular Anesthetic. J Ocul Pharmacol Ther. 2022 Sep;38(7):481-488. doi: 10.1089/jop.2022.0026. Epub 2022 Jul 18. PMID 35852839